CLINICAL TRIAL: NCT03948256
Title: Danish RAndomized Trial of External Ventricular Drainage Cessation IN Aneurysmal Subarachnoid Haemorrhage (DRAIN)
Brief Title: Danish RAndomized Trial of External Ventricular Drainage Cessation IN Aneurysmal Subarachnoid Haemorrhage
Acronym: DRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tiit Mathiesen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18054954
Record Dates: First submitted 2019-04-04; First posted 2019-05-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Hydrocephalus
Keywords: External ventricular drain; Weaning; Closure; Controlled trial; Randomised trial; Outcome assessment blinded
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hydrocephalus

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention with two arms with different time course it is not possible to mask patients nor investigators or care providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control intervention (Active Comparator): Prompt closure, based on best available scientific data
  Interventions: Procedure: Control intervention
- Experimental intervention (Experimental): Gradual weaning, based on best available scientific data
  Interventions: Procedure: Experimental intervention

INTERVENTIONS:
Procedure: Control intervention — Prompt closure of EVD with subsequent observation period
  Other Names: Prompt closure
  Arms: Control intervention
Procedure: Experimental intervention — Gradual weaning of EVD with 5 cmH2O increase in drainage resistance daily until complete closure with subsequent observation period
  Other Names: Gradual weaning
  Arms: Experimental intervention

SUMMARY:
The DRAIN trial is an international multi-centre, 1:1 randomised, parallel-group, superiority clinical trial investigating gradual weaning vs. prompt closure of external ventricular drainage in patients with hydrocephalus following aSAH.

The primary objective is to investigate the beneficial and harmful effects of gradual weaning versus prompt closure of EVD treatment in patients with aSAH.

ELIGIBILITY:
Inclusion criteria

* >= 18 years of age
* Diagnosis of aneurysmal subarachnoid haemorrhage (aSAH)
* External ventricular drain (EVD) for >= 6 days
* Drain output of =< 220 mL on day of randomisation
* Drain resistance of 10 or 15 cm H2O
* Stable or improving Glasgow Coma Scale (GCS) >= 9 during the last 24 hours
* Signed informed consent (from patient or next-of-kin)

Exclusion criteria

* None-tolerability of an increase of resistance to 10 cm H2O due to clinical deterioration or an increase in ICP
* Severe pre-existing (physical or mental) disability or severe co-morbidity that would lead to poor outcome even if the patient made a full recovery from the aSAH
* Life expectancy shorter than 48 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
VP-shunt implantation, all-cause mortality, or EVD-related infection. | 6 months after ictus
  The primary outcome is a composite outcome of VP-shunt implantation, all-cause mortality, and EVD-related infection.

SECONDARY OUTCOMES:
Number of serious adverse events (SAE) not including death | 6 months after ictus
  Number of serious adverse events (SAE) not including death as defined according to International Conference of Harmonization of Good Clinical Practice (ICH-GCP) at 6 months (count outcome)
Health-related quality of life (EQ-5D-5L) | 6 months after ictus
  Health-related quality of life (EQ-5D-5L) at 6 months with the primary assessment being self- assessment of own health (EQ VAS; 0 to 100 point scale, 100 being the best possible outcome)) (continuous outcome)

OTHER OUTCOMES:
Functional outcome according to modified Rankin Scale | 6 months after ictus
  Functional outcome according to mRS at 6 months, (1-6 scale, 1 being the best possible outcome)) (ordered categorical outcome)
The remaining dimensions of EQ-5D-5L | 6 months after ictus
  The remaining dimensions of EQ-5D-5L (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) at 6 months (1-5 levels, 1 being the best possible outcome) (count outcome)
Fatigue Severity Scale (FSS) | 6 months after ictus
  Fatigue Severity Scale (FSS) at 6 months (1-7 scale, 1 being the best possible outcome) (ordered categorical outcome)
Glasgow Outcome Scale Extended (GOSE) | 6 months after ictus
  Glasgow Outcome Scale Extended (GOSE) at 6 months (1-8 scale, 8 being the best possible outcome) (ordered categorical outcome)
Reason for failure of EVD cessation | At time of failure (assessed up to 6 months)
  Reason for failure of EVD cessation (ICP elevation, drop in GCS by 2 points or more, and/or clinical deterioration)
Glasgow Coma Score (GCS) on discharge from the Neuro Intensive Care Unit and Neurosurgical department (3-15 scale, 15 being the best possible outcome) | At time of discharge (assessed up to 6 months)
  Glasgow Coma Score (GCS) on discharge from the Neuro Intensive Care Unit and Neurosurgical department (3-15 scale, 15 being the best possible outcome)
Length of stay in Neuro Intensive Care Unit and hospital | At time of discharge (assessed up to 6 months)
  Length of stay in Neuro Intensive Care Unit and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Tiit I Mathiesen, DMSc, Principal Investigator — Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet
Locations (4):
- Denmark (2):
  - Department of Neurosurgery, Odense University Hospital, Odense, Region Syd
  - Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet, Copenhagen
- Norway (2):
  - Department of Neurosurgery, Oslo University Hospital, Oslo
  - Department of Neurosurgery, University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No
Data wille be available upon reasonable request and only after approval from local authorities and involving parties.

REFERENCES:
- [Derived] Capion T, Lilja-Cyron A, Juhler M, Moller K, Sorteberg A, Ronning PA, Poulsen FR, Wismann J, Schack AE, Ravlo C, Isaksen J, Lindschou J, Gluud C, Mathiesen T, Olsen MH. Prompt closure versus gradual weaning of external ventricular drain for hydrocephalus following aneurysmal subarachnoid haemorrhage: a statistical analysis plan for the DRAIN randomised clinical trial. Trials. 2024 Jul 15;25(1):479. doi: 10.1186/s13063-024-08305-4. PMID 39010208
- [Derived] Capion T, Lilja-Cyron A, Olsen MH, Juhler M, Moller K, Sorteberg A, Ronning PA, Poulsen FR, Wismann J, Ravlo C, Isaksen J, Lindschou J, Gluud C, Mathiesen T. Prompt closure versus gradual weaning of external ventricular drainage for hydrocephalus following aneurysmal subarachnoid haemorrhage: Protocol for the DRAIN randomised clinical trial. Acta Anaesthesiol Scand. 2023 Sep;67(8):1121-1127. doi: 10.1111/aas.14263. Epub 2023 May 10. PMID 37165711